CLINICAL TRIAL: NCT01440933
Title: Efficacy of Sugammadex for the Reversal of Moderate and Deep Rocuronium Induced Neuromuscular Block in Patients Pretreated With Magnesium Sulphate
Brief Title: Efficacy of Sugammadex in Magnesium Pretreated Patients
Acronym: MagSug
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Christoph Czarnetzki, Responsable Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER 10-093
Record Dates: First submitted 2011-09-08; First posted 2011-09-27 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Neuromuscular Block
Keywords: sugammadex; rocuronium; magnesiumsulphate; neuromuscular monitoring
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesiumsulphate (Active Comparator)
  Interventions: Drug: Magnesium Sulfate
- Physiologic saline (Placebo Comparator)
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Magnesium Sulfate — 1ml/kg of the study solution containing 60 mg/ml of magnesium sulphate are given intravenously over 15 minutes in the conscious patient. After anaesthesia induction and calibration of neuromuscular monitoring (TOF Watch SX - acceleromyography) 0,6 mg/kg of rocuronium is given intravenously. After recovery of the neuromuscular block to a posttetanic count of 2 (deep neuromuscular block) (PTC 2) or reappearance of 2 twitches of the Train of four (superficial neuromuscular block) 4 mg/kg (deep neuromuscular block) or 2 mg/kg (superficial neuromuscular block) of Sugammadex are given intravenously.
  Arms: Magnesiumsulphate
Drug: Placebo comparator — 1ml/kg of the study solution containing physiologic saline are given intravenously over 15 minutes in the conscious patient. After anaesthesia induction and calibration of neuromuscular monitoring (TOF Watch SX - acceleromyography) 0,6 mg/kg of rocuronium is given intravenously. After recovery of the neuromuscular block to a posttetanic count of 2 (deep neuromuscular block) (PTC 2) or reappearance of 2 twitches of the Train of four (superficial neuromuscular block) 4 mg/kg (deep neuromuscular block) or 2 mg/kg (superficial neuromuscular block) of Sugammadex are given intravenously.
  Arms: Physiologic saline

SUMMARY:
Sugammadex is a new reversal agent for neuromuscular blockers (curare). It encapsulates the curare molecule and terminates immediately its action. The recommended dose is 2 mg/kg for a slight neuromuscular block and 4 mg/kg for a profound neuromuscular block. Magnesium sulphate is frequently used in perioperative medicine and it is known to reinforce the neuromuscular block induced for instance by rocuronium. The researchers want to investigate, whether higher doses of sugammadex must be given to antagonize the neuromuscular block induced by rocuronium in patients who received magnesium sulphate.

DETAILED DESCRIPTION:
Neuromuscular blocking agents (NMBAs) are frequently used in anaesthesia and intensive care medicine for tracheal intubation, artificial ventilation, and continued muscle relaxation during surgical interventions. Postoperative residual curarisation is associated with an increased risk of postoperative complications and morbidity. Consequently, adequate reversal of neuromuscular block after surgery is of great importance.

Cholinesterase inhibitors have been widely used as reversal agents. They increase the amount of acetycholine at the neuromuscular junction, which then competes with the NMBA to restore muscle function. Cholinesterase inhibitors have, however, a number of limitations. They antagonise the neuromuscular block slowly and are only effective when partial spontaneous recovery has already occurred. These agents are also associated with a relatively high incidence of cholinergic adverse reactions, including bradycardia, arrhythmia, salivation, and bronchoconstriction.

Sugammadex, a modified gamma cyclodextrin, is a selective binding agent specifically designed to encapsulate steroidal NMBAs such as rocuronium. It causes a rapid and complete reversal of neuromuscular blockade by preventing directly rocuronium to react on the neuromuscular receptor.

Dose-finding studies have suggested that sugammadex 2 mg kg-1 was needed for the reversal of a moderate neuromuscular block (reappearance of T2), and that doses ≥4 mg kg-1 were needed for the reversal of a profound block (1 to 2 post-tetanic counts). The median time for the recovery of a moderate neuromuscular block to a T4/T1 ratio of 0.9 (which is considered clinically safe) is around two minutes, and of a profound neuromuscular block is about three minutes.

Magnesium is sometimes used in perioperative medicine, for instance, to prevent seizures in parturients with pre-eclampsia. Magnesium has an impact on neuromuscular transmission. It reduces the amount of acetylcholine that is released at the motor nerve terminal, by decreasing the calcium conductance of presynaptic voltage-dependent calcium channels. After pre-treatment with a clinically relevant dose of magnesium sulphate (MgSO4), an increased speed of onset and a prolongation of the recovery period of the neuromuscular blockade have been observed with standard intubation doses of atracurium, vecuronium, and rocuronium. With rocuronium, for instance, the investigators recorded a shortening of the speed of onset of the neuromuscular block by about 35% but at the expense of a prolongation of the recovery period by about 25%. It has been shown that the interaction between magnesium and rocuronium may become relevant in specific clinical situations.

The clinically relevant interaction between MgSO4 and rocuronium begs the question as to whether in a patient who has received MgSO4, the efficacy of sugammadex to reverse a rocuronium-induced block may be affected. Indeed, animal studies have indicated that significantly higher doses of sugammadex might be needed to reverse a rocuronium-induced neuromuscular block after magnesium pretreatment.

The aim of this study is to test the hypothesis that the established doses of sugammadex for the fast and safe reversal of a moderate and a profound rocuronium-induced neuromuscular block are inadequate in patients who have received MgSO4. The investigators hypothesize that in subjects who received magnesium pretreatment, the time to reverse a moderate and a deep neuromuscular block (induced by a single intubation dose of rocuronium) with standard doses of sugammadex (2 and 4 mg kg-1, respectively) is prolonged by ≥ 50% and that the dose response curves will be displaced to the right (i.e. higher doses of sugammedex will be necessary to achieve the same speed of action as in patients who are not exposed to magnesium.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to 60 years, male.
* American Society of Anesthesiology [ASA] status I or II.
* Able to read and understand the information sheet and to sign and date the consent form.
* Scheduled for elective surgery lasting at least 60 minutes under general anaesthesia requiring neuromuscular relaxation using rocuronium bromide for endotracheal intubation.

Exclusion Criteria:

* A history of allergy or hypersensitivity to rocuronium, sugammadex or magnesium
* Neuromuscular disease.
* Preoperative medications known to influence neuromuscular function (for instance, certain antibiotics [aminoglycosides] and anticonvulsants [phenytoine]).
* Electrolyte abnormalities (for instance, hypermagnaesemia).
* Hepatic dysfunction (i.e bilirubin <1.5 upper limit normal (ULN), alanine aminotransferase (ALT) <2.5 x ULN, aspartate aminotransferase (AST) <2.5 x ULN)
* Renal insufficiency (i.e. Creatinine <1.5 x ULN, creatinine clearance <30ml/minute).
* Atrioventricular heart block
* Patients with magnesium treatment
* Patients with a body mass index <19 or >28 kg m-2.
* Pregnant, or intending to become pregnant, women.
* Breastfeeding women.
* Expected difficult intubation or mask ventilation.
* Patient having participated in any clinical trial within 30 days, inclusive, of signing the informed consent form of the current trial.
* Patients needing continuous or repeat rocuronium administration for surgical reasons.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Time from start administration of sugammadex to recovery T4/T1 ratio to 0.9 | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  Neuromuscular function will be assessed by acceleromyography of the adductor pollicis with a TOF-Watch SX® monitor (Organon Oss, The Netherlands). After induction of anesthesia and loss of consciousness, the acceleromyograph will be calibrated using the implemented TOF-Watch SX® calibration mode 2. Train-of-four (TOF) stimulation will be used (supramaximal square wave impulse of 200 µs duration, four stimuli at two Hz, 15 seconds interval). The units of measurement are seconds and minutes. Measurement will be continued until a TOF ration of 1.0 is reached.

SECONDARY OUTCOMES:
Time from start administration of sugammadex to recovery T4/T1 ratio to 0.7 | Participants will be followed for the duration of hospital stay, an expected average of 2 days
  Neuromuscular function will be assessed by acceleromyography of the adductor pollicis with a TOF-Watch SX® monitor (Organon Oss, The Netherlands). After induction of anesthesia and loss of consciousness, the acceleromyograph will be calibrated using the implemented TOF-Watch SX® calibration mode 2. Train-of-four (TOF) stimulation will be used (supramaximal square wave impulse of 200 µs duration, four stimuli at two Hz, 15 seconds interval). The units of measurement are seconds and minutes. Measurement will be continued until a TOF ration of 1.0 is reached.
Time from start administration of sugammadex to recovery T4/T1 ratio to 0.8. | SParticipants will be followed for the duration of hospital stay, an expected average of 2 days
  Neuromuscular function will be assessed by acceleromyography of the adductor pollicis with a TOF-Watch SX® monitor (Organon Oss, The Netherlands). After induction of anesthesia and loss of consciousness, the acceleromyograph will be calibrated using the implemented TOF-Watch SX® calibration mode 2. Train-of-four (TOF) stimulation will be used (supramaximal square wave impulse of 200 µs duration, four stimuli at two Hz, 15 seconds interval). The units of measurement are seconds and minutes. Measurement will be continued until a TOF ration of 1.0 is reached.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Czarnetzki, MD, MBA, Principal Investigator — Universital Hospitals of Geneva; Martin R Tramer, MD, Dphil, Study Chair — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland